CLINICAL TRIAL: NCT05371288
Title: The Role of Glutathione Deficiency and MSIDS Variables in Long COVID-19
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No longer studying long COVID
Sponsor: University of California, Irvine (Other)
Collaborators: Hudson Valley Healing Arts Center (Unknown)
Responsible Party: Principal Investigator, Alpesh N Amin, Principal Investigator, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCR-21-128
Record Dates: First submitted 2022-04-08; First posted 2022-05-12 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
Keywords: Covid-19 Long-Haul
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Acetylcysteine; Thioctic Acid; Glutathione

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- No Multivitamin and Magnesium (Experimental): Subjects randomized into Group A will take the following amount for 28 days
  * 4 capsules of NAC (600mg each) once in the morning and once in the evening
  * 1 tablet (600mg) of Alamax CR once in the morning and once in the evening
  * 8 capsules (250 mg each) of liposomal GSH in the morning and in the evening
  Interventions: Drug: NAC (N-acetyl cysteine), Alpha lipoic acid (ALA), liposomal glutathione (GSH)
- Multivitamin and Magnesium (Active Comparator): Subjects randomized into Group B will be taking a multivitamin and magnesium for 14 days. Afterwards, they will take the following for 14 days.
  * 4 capsules of NAC (600mg each) once in the morning and once in the evening
  * 1 tablet (600mg) of Alamax CR once in the morning and once in the evening
  * 8 capsules (250 mg each) of liposomal GSH in the morning and in the evening
  Interventions: Drug: NAC (N-acetyl cysteine), Alpha lipoic acid (ALA), liposomal glutathione (GSH)

INTERVENTIONS:
Drug: NAC (N-acetyl cysteine), Alpha lipoic acid (ALA), liposomal glutathione (GSH) — Nutritional supplements hypothesized to help reverse some of the COVID long-haul symptoms.

SUMMARY:
The purpose of this research study is to assess if glutathione, along with NAC (N-acetyl cysteine) and Alpha lipoic acid (ALA), can help reverse some of the COVID long-haul symptoms.Subjects will be randomized in to one of two groups. Depending on the group they are randomized in to, subjects will be taking either a combination of NAC, Alamax CR, and liposomal GSH or the same three nutritional supplements with a multivitamin and magnesium. Regardless of the group, subjects will be asked questions to assess their COVID symptoms, physical and mental health status. They will also be asked to take blood samples.

ELIGIBILITY:
Inclusion Criteria:

• Patients with positive COVID testing (AB, RT PCR) and mild-severe symptoms based on COVID symptom list

Exclusion Criteria:

• History of a severe sulfa sensitivity (i.e., anaphylaxis, Stevens Johnson Syndrome), allergy to meat products and/or gelatin (alpha gal allergy) and/or a history of an allergic or adverse reaction to NAC, alpha lipoic acid and/or GSH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Assess Changes in Symptoms of Post-Acute Sequelae of COVID (PASC) | Symptoms will be evaluated at 2 weeks, 1-, 2-, 3- and 4 months post therapy
  With the goal of reversing symptoms of Post-Acute Sequelae of COVID, this outcome measure aims to evaluate changes in symptoms before and after therapy, and determining which, if any symptoms are improved in each arm of the trial.
Change in Quality of Life Using SF-36 Survey | Will be evaluated at 2 weeks, 1-, 2-, 3- and 4 months post therapy
  The SF-36 survey is a multipurpose, short-form health survey with 36 questions to evaluate health-related Quality of Life . It yields an eight-scale profile of scores as well as physical and mental health summary measures. It is a generic measure, as opposed to one that targets a specific age, disease, or treatment group.
COVID Severity of Symptoms Questionnaire | Day 15, 28, end of months 2, 3, 4
  This will evaluate the changes in the severity of symptoms over time with treatment.
Change in Time to Clinical Recovery (TTCR) | Day 15 and 28 (month 1), and at the end of months 2, 3 and 4
  Starting on day one of subjects' treatment, subjects will be asked if symptoms have improved or worsened, and the time it took for symptoms to change since their last treatment: (0 [no change], +1 [improved within 7 days], + 2 [improved within 14 days], +3 [improved within 28 days] + 4 [symptom resolved]; - 1 [worsened within 7 days], -2 [worsened within 14 days], - 3 [worsened within 28 days], - 4 [debilitating last 28 days]

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No